CLINICAL TRIAL: NCT02865811
Title: A Phase II Study of Pembrolizumab Combined With Pegylated Liposomal Doxorubicin (PLD) For Recurrent Platinum Resistant Ovarian, Fallopian Tube Or Peritoneal Cancer
Brief Title: Pembrolizumab Combined With PLD For Recurrent Platinum Resistant Ovarian, Fallopian Tube Or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ursula A. Matulonis, MD, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-257
Record Dates: First submitted 2016-08-10; First posted 2016-08-12 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — pembrolizumab; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab in Combination With PLD (Experimental): A safety lead in with 6 patients will be studied prior the start of the treatment.
  * If 2 out of the first 6 patients develop a dose limiting toxicity (DLT), the dose of PLD will be reduced.
  * If no more than 1 patient of the first 6 patients has evidence of dose limiting toxicities, the dose level will be considered the maximum tolerated dose (MTD)
  * Pegylated Liposomal Doxorubicin (PLD) pre-determine dosage will be administered every 4 weeks via IV
  * Pembrolizumab will be administered as a 30 min IV infusion every 3 weeks at a pre-determine dosage
  Interventions: Drug: Pembrolizumab; Drug: Pegylated Liposomal Doxorubicin (PLD)

INTERVENTIONS:
Drug: Pembrolizumab — Please see "Arms" for description.
  Other Names: Keytruda
Drug: Pegylated Liposomal Doxorubicin (PLD) — Please see "Arms" for description.

SUMMARY:
This research study is studying the combination of Pegylated Liposomal Doxorubicin (PLD) and Pembrolizumab as a possible treatment for Recurrent Ovarian, Fallopian Tube or Peritoneal Cancer that is resistant to platinum therapy.

The following interventions will be used in this study:

* Pegylated liposomal doxorubicin (PLD)
* Pembrolizumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The investigators are looking to see if combining the standard therapy, PLD, and the study drug, Pembrolizumab, will be better than PLD alone. Pembrolizumab is a drug called a monoclonal antibody. Pembrolizumab blocks and interferes with a protein called PD-1; PD-1 can help the cancer cell evade the immune system, and thereby blocking PD-1 may help the immune system recognize and kill cancer cells.

This will be the first time this combination will be tested for participants with Ovarian, Fallopian Tube or Peritoneal Cancer. Therefore, a group of 6 participants will be treated in a "safety lead in" portion of the trial. This lead in will determine the safest dose of PLD when given in combination with the study drug Pembrolizumab. These 6 participants will be treated with Pembrolizumab and PLD at the FDA approved dose to see if the combination is well tolerated or too severe. If the combination is well tolerated, 20 additional participants will be added. If the side effects are too severe, the dose of PLD will be lowered.

The FDA (the U.S. Food and Drug Administration) has approved PLD as a treatment option for this disease, but has not approved Pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1 criteria.
* Have a histologically confirmed diagnosis of epithelial ovarian cancer, fallopian tube or peritoneal cancer. All histologies of epithelial ovarian cancer are eligible except for carcinosarcomas.
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound. This initial treatment may have included intraperitoneal therapy, consolidation, biologic/targeted (non-cytotoxic) agents (e.g., bevacizumab) or extended therapy administered after surgical or non-surgical assessment.
* Patients must have platinum resistant cancer with a platinum free interval of < 6 months. Progression after last platinum is based on investigator assessment.
* Patients are allowed to receive, but are not required to receive, up to two additional cytotoxic regimens for management of recurrent or persistent disease, with no more than 1 non-platinum, non-taxane regimen.
* Patients are allowed to receive, but are not required to receive, biologic/targeted (non-cytotoxic) therapy as part of their primary treatment regimen. For the purposes of this study, Poly (ADP-ribose) polymerase (PARP) inhibitors will be considered "cytotoxic." Patients are allowed to receive, but are not required to receive, PARP inhibitors for management of primary or recurrent/persistent disease (either alone or in combination with cytotoxic chemotherapy). Single agent hormonal therapies will not be counted as a line of treatment.
* Have adequate tissue from an archived specimen of ovarian cancer (between 10 to 15 slides of unstained tumor).
* Have a performance status of 0 or 1 on the ECOG Performance Scale (Appendix A).
* Demonstrate adequate organ function as defined in Table 1, all screening labs must be performed within 10 days of treatment initiation.

Table 1 Adequate Organ Function Laboratory Values

System Laboratory Value

* Hematological

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
* Renal

  * Serum creatinine OR
  * Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for participant with creatinine levels > 1.5 X institutional ULN
* Hepatic

  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for participants with liver metastases
  * Albumin >2.5 mg/dL
* Coagulation

  * International Normalized Ratio (INR) or Prothrombin Time (PT)
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.
* Female participants of childbearing potential must have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Patients cannot have primary platinum refractory cancer, i.e. documented cancer progression while receiving platinum or within one month of receipt of a platinum based regimen.
* Has received a prior anthracycline chemotherapy either for ovarian cancer treatment or another previous malignancy.
* Left ventricular ejection fraction (LVEF) defined by multigated acquisition (MUGA) or echocardiogram which is below the institutional lower limit of normal prior to starting study treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients and/or liposomal doxorubicin.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Participants with < Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If participant underwent major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. In addition, patients cannot have been diagnosed with another malignancy within 3 years of starting treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include clinically active and significant carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2022-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Matulonis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Northwell Hospital Monter Cancer Center, Lake Success, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee EK, Xiong N, Cheng SC, Barry WT, Penson RT, Konstantinopoulos PA, Hoffman MA, Horowitz N, Dizon DS, Stover EH, Wright AA, Campos SM, Krasner C, Morrissey S, Whalen C, Quinn R, Matulonis UA, Liu JF. Combined pembrolizumab and pegylated liposomal doxorubicin in platinum resistant ovarian cancer: A phase 2 clinical trial. Gynecol Oncol. 2020 Oct;159(1):72-78. doi: 10.1016/j.ygyno.2020.07.028. Epub 2020 Aug 6. PMID 32771276

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab in Combination With PLD: A safety lead in with 6 patients will be studied prior the start of the treatment.
  * If 2 out of the first 6 patients develop a dose limiting toxicity (DLT), the dose of PLD will be reduced.
  * If no more than 1 patient of the first 6 patients has evidence of dose limiting toxicities, the dose level will be considered the maximum tolerated dose (MTD)
  * Pegylated Liposomal Doxorubicin (PLD) pre-determine dosage will be administered every 4 weeks via IV
  * Pembrolizumab will be administered as a 30 min IV infusion every 3 weeks at a pre-determine dosag
Period: Overall Study
Arm/Group | Pembrolizumab in Combination With PLD
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab in Combination With PLD
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (11.3)
Age, Customized [Median (Full Range); unit: years] | 60.0 [28.3 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 1
  Unknown or Not Reported | 0
Stage at Initial Diagnosis [Count of Participants; unit: Participants]
  Stage I | 2
  Stage II | 1
  Stage III | 12
  Stage IV | 10
  Missing | 1
Differentiation (Grade) [Count of Participants; unit: Participants]
  Well Differentiated | 1
  Moderately Differentiated | 1
  Poorly Differentiated | 21
  Missing | 3
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma, not further specified | 1
  Serous | 20
  Clear Cell | 2
  Mucinous | 2
  Mixed serous/mucinous | 1
ECOG Performance Status [Count of Participants; unit: Participants]
  0- Fully Active | 16
  1- Restricted | 10
# of Prior Lines [Count of Participants; unit: Participants]
  1 | 10
  2 | 10
  3 | 6
Platinum Free Interval (PFI) [Count of Participants; unit: Participants]
  <3 Months | 7
  3-6 Months | 19

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate [CBR]
Description: The primary objective was to determine the CBR (complete response [CR] + partial response [PR] + stable disease [SD] >/= 24 weeks) of the combination of pembrolizumab and PLD.
Time Frame: 24 Weeks
Population: Of the 26 patients enrolled, 23 patients were evaluable for objective response by RECIST.
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab in Combination With PLD: A safety lead in with 6 patients will be studied prior the start of the treatment.
  * If 2 out of the first 6 patients develop a dose limiting toxicity (DLT), the dose of PLD will be reduced.
  * If no more than 1 patient of the first 6 patients has evidence of dose limiting toxicities, the dose level will be considered the maximum tolerated dose (MTD)
  * Pegylated Liposomal Doxorubicin (PLD) pre-determine dosage will be administered every 4 weeks via IV
  * Pembrolizumab will be administered as a 30 min IV infusion every 3 weeks at a pre-determine dosage
  Pembrolizumab: Please see "Arms" for description.
  Pegylated Liposomal Doxorubicin (PLD): Please see "Arms" for description.
Arm/Group | Pembrolizumab in Combination With PLD
Number analyzed (Participants) | 23
Participants | 12

2. Secondary Outcome: Safety of the Combination of Pembrolizumab/PLD
Description: Safety is measured by any dose limiting toxicity experienced within the safety lead in group of 6 patients. If 2 out of the first 6 patients develop a DLT, the dose of PLD will be reduced to 30 mg/m2. If no more than 1 patient of the first 6 patients has evidence of dose limiting toxicities, the dose level will be considered the maximum tolerated dose (MTD), an additional 20 patients will be enrolled to complete the phase II study.
Time Frame: 24 weeks
Population: 6 patients were included in the safety lead-in group
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab in Combination With PLD
Number analyzed (Participants) | 6
Participants | 1

3. Secondary Outcome: Overall Response Rate [ORR]
Description: A secondary objective was to determine the Overall Response Rate [ORR] of the combination of pembrolizumab and PLD as defined by the number of participants achieving a partial response [PR] or complete response [CR].
Time Frame: 24 months
Population: Of the 26 patients enrolled, 23 patients were evaluable for objective response by RECIST.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab in Combination With PLD
Number analyzed (Participants) | 23
Participants
  Partial Response | 5
  Complete Reponse | 1

4. Secondary Outcome: Duration of Response [DOR]
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation).
Time Frame: 24 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab in Combination With PLD
Number analyzed (Participants) | 26
months | 10.58 [2.56 to NA] — There are not enough events to estimate the upper confidence limit for the duration of response, therefore the upper limit of the response curve hasn't reached 50% probability which is the median line.

5. Secondary Outcome: Progression-Free Survival [PFS]
Description: Progression-Free Survival is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without progression are censored at date of last disease evaluation.
Time Frame: 24 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab in Combination With PLD
Number analyzed (Participants) | 26
months
  Progression events defined by RECIST 1.1 | 8.1 [1.7 to 14.7]
  Progression events defined by RECIST 1.1 and clinical progression | 5.6 [1.7 to 10.1]

6. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Time Frame: 24 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab in Combination With PLD
Number analyzed (Participants) | 26
months | 18.3 [9.4 to 31.5]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected weekly throughout study participation for all patients, and for 4 weeks after treatment completion.
Description: Expedited reporting applied to any medical event equivalent to an unexpected grade 2 or 3 with a possible, probable or definite attribution, both expected (unless listed in the protocol as not requiring expedited reporting) and unexpected grade 4 toxicities, and grade 5 (death) regardless of study phase or attribution.
Arm/Group | Pembrolizumab in Combination With PLD
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 3/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab in Combination With PLD (N=26)
Alanine aminotransferase increased (Investigations) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (2)
Seizure (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab in Combination With PLD (N=26)
Fatigue (General disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10
Anemia (Blood and lymphatic system disorders) | 9
Constipation (Gastrointestinal disorders) | 8
Aspartate aminotransferase increased (Investigations) | 8
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 8
Diarrhea (General disorders) | 7
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 7
Infections and infestations - Other, specify (Infections and infestations) | 7
Hyponatremia (Metabolism and nutrition disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 5
Fever (General disorders) | 5
Pain (General disorders) | 5
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 5
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 5
Mucositis oral (Gastrointestinal disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Ascites (Gastrointestinal disorders) | 4
Small intestinal obstruction (Gastrointestinal disorders) | 4
Urinary tract infection (Infections and infestations) | 4
Hypothyroidism (Endocrine disorders) | 3
Oral pain (Gastrointestinal disorders) | 3
Infusion related reaction (General disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Upper respiratory infection (Infections and infestations) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Fecal incontinence (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 2
Skin infection (Infections and infestations) | 2
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Urinary urgency (Renal and urinary disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Mucosal infection (Infections and infestations) | 2
Pneumonitis (Reproductive system and breast disorders) | 2
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Dry eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroparesis (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Oral dysesthesia (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Sinusitis (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 1
Weight loss (Investigations) | 1
Dysgeusia (Nervous system disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Urostomy obstruction (Injury, poisoning and procedural complications) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Sepsis (Infections and infestations) | 1
Seizure (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT02865811/Prot_SAP_000.pdf